CLINICAL TRIAL: NCT00323180
Title: Investigation of Protein Biomarkers of Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution and no subjects enrolled and this is not a clinical trial.
Sponsor: University of New Mexico (Other)
Responsible Party: Marco Bisoffi; Principal Investigator, Universtiy of New Mexico
Other Study IDs: HRRC 03-376
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is looking at biomarkers in prostate cancer.

DETAILED DESCRIPTION:
1. To establish primary culture of epithelial cells isolated from prostatectomy samples
2. To study biomarkers in prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bisoffi, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States